CLINICAL TRIAL: NCT05796076
Title: Virtual Reality Intervention on Anxiety and Pain Among Adult Patients Ubdergoing an Awake Minor Suture: A Pilot Randomized Controlled Trial
Brief Title: Virtual Reality to Reduce Anxiety and Pain During Suturing Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Collaborators: Tung Wah College (Other)
Responsible Party: Principal Investigator, Ko Shuk Yee, Advanced Practice Nurse, Tuen Mun Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NTWC/REC/22003
Record Dates: First submitted 2023-03-06; First posted 2023-04-03 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Suture
Keywords: Anxiety; Pain; Virtual reality; Suturing
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Intervention and control group
Masking Description: Investigator will not be involved the recruitment and data collection. Outcome assessor will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control group (Other): Participants in the control group will be received standard care
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — Participants in the intervention group will be received VR during the suturing procedure. Virtual reality is a three dimensions of width, height and depth that is generated digitally in a computer-generated environment that allows a user to interact with it 16.

SUMMARY:
Background: In emergency departments, suturing is a common procedure but often causes anxiety and pain. Virtual reality (VR) intervention has been reported as a relaxing measure.

Objective: The study aims to examine the effects of VR intervention on anxiety, pain, physiological parameters, local anaesthesia requirements and satisfaction in Chinese adult patients undergoing wound closure in emergency departments in Hong Kong

Hypothesis:VR can alleviate anxiety and pain experienced by Chinese adult patients undergoing wound-closure procedures, the intervention can decrease extra local anesthesia requirements and physiological parameters during the procedures, and the intervention can significantly increase satisfaction during wound-closure procedures.

DETAILED DESCRIPTION:
Suturing is one of the most common procedure in the emergency department, however, it often provokes anxiety and pain. 1-2 Failure to manage patients' anxiety and pain during wound closure can cause difficulties for health care providers to complete the procedures and reduce the success rates. 3 Experience of anxiety and pain may also increase the need for medication, reduce patients' satisfaction rate and cause negative physiological parameters such as increased blood pressure and heart rate. 4-5.

Traditionally, nonpharmacological intervention such as listening to music, chatting, and guided imagery is applied to reduce patient's anxiety and pain. However these measures fail to provide patients with significant distraction because patients would inevitably see the procedure that causes considerable distress during the procedure. Thus, the development of further strategies to provide a significant distraction to alleviate patients' anxiety and pain during suturing is warranted.

With advanced technologies, virtual reality (VR) provides significant distraction. Clinical trials indicate that use of VR achieved a statistically significant decrease in anxiety and pain in different operations such as hand 6, lipoma incision 7, Gynecology 8, and debridement 9. However, only a handful of studies conducted among adult patient with ambulatory laceration repairing examined the effectiveness of VR in anxiety and pain. To the best of our knowledge, no study specifically focus on the effects of VR on anxiety and pain in Chinese adult patients undergoing an awake suture in emergency room in Hong Kong. Eighty participants will be assigned to the experimental group or to the control group by randomization.

After written informed consent will be obtained from patients, the baseline data (T0) will be obtained from the participants including sociodemographic, anxiety, blood pressure, and pulse rate. Subsequently, randomization is conducted. Throughout the procedure (T1), the additional medication requirements and physiological parameters will be recorded. The anxiety, pain and satisfaction and physiological parameters will also be recorded after the procedure. Data will be analyzed using IBM SPSS 23.0. Descriptive statistics, including frequency, percentage, mean and standard deviation will be used to describe the data. Chi-square tests compare categorical variables, and independent t-tests compare continuous variables. Generalized Estimation Equation will be used to examine the effectiveness of the VR intervention versus the control group will be evaluated by comparing the study outcomes. Two-tailed tests will be used with a significant level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Conscious, oriented
2. Adult patient (age between 18 and 65 years) with scheduled to receive an awake minor suture
3. Ability to communicate in Chinese, and read and write Chinese language
4. Hemodynamic stability as evidenced by blood pressure between 90 to 140 mmHg systolic and 60 to 90 mmHg diastolic before the procedure

Exclusion Criteria:

1. Have visual, hearing or cognitive impairment
2. History of senile dementia, seizure disorder, motion sickness, psychiatric disorders as indicated in medical record
3. Have injury or infection above the neck
4. Known to be on contact precaution

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Anxiety | Baseline, and 5 minutes after the completion of the procedure
  The Chinese version of the State Trait Anxiety scale is used to measure anxiety levels of the patients. It contains two separate scales for state and trait anxiety.
  The first part (state anxiety) evaluates a transitory emotional state that is influenced by intense emotional situations and varies in intensity over time. The second part (trait anxiety) demonstrates a relatively stable anxious tendency and is not significantly influenced by emotionally intense situations. Each item is rated on a 4-point Likert scale, with total scores from 20 to 80. The high the score indicates the high a higher level of anxiety. The STAI-C is validated in Hong Kong and is found to have a high degree of internal consistency (Alpha = 0.9). Participants will be required to complete the state form at 5 minutes after the completion of the procedure in this study 10-12

SECONDARY OUTCOMES:
Pain Level | During the procedure
  Pain is measured by visual analogue scales (VAS). VAS is a commonly used method for quantifying pain. The scale comprises a 10cm line with terms representing the extremes of pain at either end. The patient estimates pain by placing a mark on the line. The distance from the zero point is then measured. The VAS has been shown to be a valid tool for the measurement of psychological and health variables such as pain and satisfaction which had been used in clinical studies widely 13-15.
Satisfaction level | 5 minutes after the completion of the procedure
  Satisfaction is measured by visual analogue scales (VAS). VAS is a commonly used method for quantifying pain. The scale comprises a 10cm line with terms representing the extremes of pain at either end. The patient estimates satisfaction by placing a mark on the line. The distance from the zero point is then measured. The VAS has been shown to be a valid tool for the measurement of psychological and health variables such as pain and satisfaction which had been used in clinical studies widely 13-15.
Blood pressure | Baseline, during and 5 minutes after the completion of the procedure
  A standard blood pressure monitor is used to measure patients' blood pressure. The blood pressure is recorded as mmHg
Pulse rate | Baseline, during and 5 minutes after the completion of the procedure
  A standard pulse oximetry is used to measure patients' pulse rate. The pulse rate is recorded as beat per minute (bpm)
Additional local analgesic requirements | During the procedure
  The frequency of extra local analgesic use (1 % Lidocaine) is recorded

CONTACTS AND LOCATIONS:
Overall Officials: KO SHUK YEE, DN, Principal Investigator — Tuen Mun Hospital
Locations (1):
- Tuen Mun Hospital-Emergency department, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
It is only a pilot study and will be modified after the pilot study. We will share it later on in the main study

REFERENCES:
- [Background] Bryl AW, Bonsu B, Johnson AL, Pommert KBJ, Hollenbach KA, Kanegaye JT. Tablet Computer as a Distraction Tool During Facial Laceration Repair: A Randomized Trial. Pediatr Emerg Care. 2021 Aug 1;37(8):e425-e430. doi: 10.1097/PEC.0000000000001626. PMID 30422942
- [Background] Ploghaus A, Narain C, Beckmann CF, Clare S, Bantick S, Wise R, Matthews PM, Rawlins JN, Tracey I. Exacerbation of pain by anxiety is associated with activity in a hippocampal network. J Neurosci. 2001 Dec 15;21(24):9896-903. doi: 10.1523/JNEUROSCI.21-24-09896.2001. PMID 11739597
- [Background] Parker SIA, Benzies KM, Hayden KA. A systematic review: effectiveness of pediatric peripheral intravenous catheterization strategies. J Adv Nurs. 2017 Jul;73(7):1570-1582. doi: 10.1111/jan.13211. Epub 2016 Dec 14. PMID 27864995
- [Background] De Oliveira GS Jr, Holl JL, McCarthy RJ, Butt ZA, Nouriel J, McCaffery K, Wolf MS. Overestimation of mortality risk and preoperative anxiety in patients undergoing elective general surgery procedures: a propensity matched analysis. Int J Surg. 2014 Dec;12(12):1473-7. doi: 10.1016/j.ijsu.2014.11.016. Epub 2014 Nov 18. PMID 25463769
- [Background] Robleda G, Sillero-Sillero A, Puig T, Gich I, Banos JE. Influence of preoperative emotional state on postoperative pain following orthopedic and trauma surgery. Rev Lat Am Enfermagem. 2014 Oct;22(5):785-91. doi: 10.1590/0104-1169.0118.2481. PMID 25493674
- [Background] Hoxhallari E, Behr IJ, Bradshaw JS, Morkos MS, Haan PS, Schaefer MC, Clarkson JHW. Virtual Reality Improves the Patient Experience during Wide-Awake Local Anesthesia No Tourniquet Hand Surgery: A Single-Blind, Randomized, Prospective Study. Plast Reconstr Surg. 2019 Aug;144(2):408-414. doi: 10.1097/PRS.0000000000005831. PMID 31348351
- [Background] Mosso Vazquez JL, Mosso Lara D, Mosso Lara JL, Miller I, Wiederhold MD, Wiederhold BK. Pain Distraction During Ambulatory Surgery: Virtual Reality and Mobile Devices. Cyberpsychol Behav Soc Netw. 2019 Jan;22(1):15-21. doi: 10.1089/cyber.2017.0714. Epub 2018 Sep 25. PMID 30256662
- [Background] Mosso Vázquez JL, Lara Vaca V, Wiederhold BK, Miller IT, Wiederhold MD. Virtual reality pain distraction during gynecological surgery - a report of 44 cases. Surgical Research Updates. 2017;5(1):12-16. doi: 10.12970/2311-9888.2017.05.
- [Background] Hoffman HG, Patterson DR, Seibel E, Soltani M, Jewett-Leahy L, Sharar SR. Virtual reality pain control during burn wound debridement in the hydrotank. Clin J Pain. 2008 May;24(4):299-304. doi: 10.1097/AJP.0b013e318164d2cc. PMID 18427228
- [Background] Spielberger CD, Gorsuch RC, Lushene RF. Manual of the State Trait Anxiety Inventory. Palo Alto, CA: Consulting psychologists Press; 1970
- [Background] Shek DTL. The factorial structure of the Chinese version of the state-trait anxiety inventory: a confirmatory factor analysis. Psychol Edu Meas. 1991;51(4):985-997. doi:10.1177/001316449105100418
- [Background] Shek DT. The Chinese version of the State-Trait Anxiety Inventory: its relationship to different measures of psychological well-being. J Clin Psychol. 1993 May;49(3):349-58. doi: 10.1002/1097-4679(199305)49:33.0.co;2-j. PMID 8315037
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Kersten P, White PJ, Tennant A. Is the pain visual analogue scale linear and responsive to change? An exploration using Rasch analysis. PLoS One. 2014 Jun 12;9(6):e99485. doi: 10.1371/journal.pone.0099485. eCollection 2014. PMID 24921952
- [Background] Bodian CA, Freedman G, Hossain S, Eisenkraft JB, Beilin Y. The visual analog scale for pain: clinical significance in postoperative patients. Anesthesiology. 2001 Dec;95(6):1356-61. doi: 10.1097/00000542-200112000-00013. PMID 11748392
- [Background] Moskaliuk J, Kimmerle J, Cress U. Virtual reality 2.0 and its application in knowledge building. In handbook of research on web 2.0, 3.0, and X. O: technologies, business and social applications. USA: IGI Global, 2010.